CLINICAL TRIAL: NCT07201649
Title: Roles of Hepatic Insufficiency, Hepatic Fibrosis, and Inorganic Pyrophosphate in the Progression of Arterial Calcifications
Acronym: PYROCALM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-PP-15
Record Dates: First submitted 2025-09-22; First posted 2025-10-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients eligible for Hepatit Transplantation (Other): Patients eligible for HT are contacted by a clinical research coordinator, and if they agree, an inclusion visit is arranged. HT takes place according to transplant availability. As soon as the patient is able to return home after HT, a visit is organised, defining the T1 period. A visit is carried out 120 days after HT and the end-of-study visit is scheduled to define the T2 period, which is the same length as the T1 period for each patient.
  Interventions: Other: a blood test and urine sample collection.

INTERVENTIONS:
Other: a blood test and urine sample collection. — The study is offered to all patients who meet the inclusion criteria during their pre-transplant assessment by the principal investigator (during an existing visit). Patients eligible for HT are contacted by a clinical research coordinator, and if they agree, an inclusion visit is arranged.

SUMMARY:
Individuals with metabolic syndrome (MetS), particularly those with type 2 diabetes (T2D), and/or metabolic dysfunction-associated steatohepatitis or MASH face an elevated risk of major cardiovascular events (MACE). We showed decrease plams level of PPi in patients with liver cirrhosis. We hypothezised that liver transplant should block AC and restore PPi plasma level.

ELIGIBILITY:
Inclusion Criteria:

* everyone requiring liver transplantation for the treatment of a chronic liver disease

Exclusion Criteria:

* MELD score >25, viral replication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2028-11-24 (Estimated); Study Completion 2029-11-24 (Estimated)

PRIMARY OUTCOMES:
hepatic transplantation reduces arterial calcification | On the 7th day after surgery
  compare the percent of patients with AC progression before and after liver tranplantation

SECONDARY OUTCOMES:
identify arterial calcification related factors | On the 7th day after surgery
  separation of patients according to AC progression (yes or no) and machine learning analysis with all relevant factors
increase of PPi plasma level after liver transplantation | at inclusion and at 3 months
  comparison of mean plasma levels before and after

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FAVRE, PhD, Principal Investigator — CRC, Néphrologie - CHU de Nice - Hôpital de l'Archet
Locations (1):
- CHU de Nice, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided